CLINICAL TRIAL: NCT04330014
Title: Factor Affecting Childhood Immunization Among Childern Below Two Years
Brief Title: Factor Affecting Childhood Immunization Among Childern.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Gamal Ahmed, assistant lecturer, Assiut University
Other Study IDs: Child Immunization
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Child Immunization
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: vaccine — affect vaccination on children

SUMMARY:
The aim of study to evaluate the factor affecting underutalization of childhood vaccination immunization among childern below two years of age.

DETAILED DESCRIPTION:
Childhood vaccination has proven to be one of the most effective public health strategies to control and prevent disease.1-5 In an effort to reduce childhood morbidity and mortality, the Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices (ACIP) issues annual recommendations and guidelines for childhood and adolescent immunizations.2,6-8 However, some parents decline or delay vaccinating their children or follow alternative immunization schedules because of medical, religious, philosophical, or socioeconomic reasons.2,3,4,5,7,9-12Health care provider-based interventions have been suggested to overcome such vaccine noncompliance, including patient counseling; improving access to vaccinations; maximizing patient office visits; offering combination vaccines; and using electronic medical records (EMRs) and practice alerts.2,3,4,7,10,11 Community- and government-based interventions to improve parent and patient adherence include public education and reminder/recall strategies, financial incentives, and providing alternative venues for vaccination.2,7.

ELIGIBILITY:
Inclusion Criteria:

* All childern in first two years of life who admmitted in hospital or out patient clinic.

Exclusion Criteria:

* : Immunodeficiency (e.g chemotherapy,long term immuno suppressive therapy, hematologic tumor).

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: childern below two years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between childern below two years who took vaccinations and those who didnot. | Baseline
  The investigators evaluate factors effect of vaccine on the child as scioeconomic status, poverty, chronic disease and residance.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, professor, Principal Investigator — Assiut University; Ismail Lotfy, professor, Principal Investigator — Assiut University

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4927017/